CLINICAL TRIAL: NCT01853397
Title: An Evaluation of the Safety and Effectiveness of Treatment of Adipose Tissue With the Liposonix System (Model 2) Using a New Treatment Method
Brief Title: Evaluation of the Treatment of Adipose Tissue With Liposonix System (Model 2) Using a New Treatment Method
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Solta Medical (Industry)
Responsible Party: Sponsor
Organization: Valeant Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13-137-LP-H
Record Dates: First submitted 2013-05-08; First posted 2013-05-15 (Estimated); Results first posted 2015-03-27 (Estimated); Last update posted 2015-04-16 (Estimated); Status verified 2015-03

CONDITIONS: Subcutaneous Adipose Tissue

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Treatment at level 1 (Experimental): Single treatment with Liposonix System (Model 2) using single pass technique at level 1 (180 J/cm2)
  Interventions: Device: Liposonix System (Model 2)
- Treatment at level 2 (Experimental): Single treatment with Liposonix System (Model 2)using the single pass technique at treatment level 2 (140 J/cm2)
  Interventions: Device: Liposonix System (Model 2)
- Treatment at level 3 (Experimental): Single treatment with Liposonix System (Model 2)using single pass technique at level 3 (120 J/cm2)
  Interventions: Device: Liposonix System (Model 2)
- Treatment with 3 passes at 60 J/cm2 (Active Comparator): Single treatment with Liposonix System (Model 2) using grid repeat technique with 3 passes at 60 J/cm2 (180 J/cm2 total fluence)
  Interventions: Device: Liposonix System (Model 2)

INTERVENTIONS:
Device: Liposonix System (Model 2)

SUMMARY:
The purpose of this study is to evaluate the safety, efficacy, and tolerability of treatment with the Liposonix System (Model 2)using a single pass technique.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 to 65 years of age
* Body Mass Index of ≤30 kg/m2
* Thickness of subcutaneous adipose tissue in the anticipated treatment area of ≥ 2.3 cm
* Subjects must agree to not alter their normal and regular diet or exercise routines during the course of the study
* Subject must understand the nature of the study and sign an IRB approved Informed Consent

Exclusion Criteria:

* Subject is pregnant
* Subject is diagnosed with coagulation disorders or are receiving anticoagulant therapy or medications or dietary supplements which impede coagulation or platelet aggregation
* Subject has diabetes or cardiovascular disease
* Subject has had prior aesthetic procedures to the region to be treated
* Subject has had previous open or laparoscopic surgery in the anticipated treatment area
* Subject is on prescription or over the counter weight reduction medication or programs, or had weight reduction procedures
* Subjects undergoing chronic steroid or immunosuppressive therapy
* Subject has cardiac pacemakers or any implantable electrical device
* Subject has a History of cancer
* Subject has sensory loss or dysesthesia in the area to be treated
* Subjects who are unable, or lack the capacity, to self consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2013-04; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Jewell, MD, Principal Investigator — Jewell Plastic Surgery Center; Ronald Wheeland, MD, Principal Investigator — Solta Medical Aesthetic Center
Locations (2):
- United States (2):
  - Solta Medical Aesthetic Center, Hayward, California
  - Jewell Plastic Surgery Center, Eugene, Oregon

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment at Level 1: Single treatment with Liposonix System (Model 2) using single pass technique at level 1 (180 J/cm2)
  Liposonix System (Model 2)
- Treatment at Level 2: Single treatment with Liposonix System (Model 2)using the single pass technique at treatment level 2 (140 J/cm2)
  Liposonix System (Model 2)
- Treatment at Level 3: Single treatment with Liposonix System (Model 2)using single pass technique at level 3 (120 J/cm2)
  Liposonix System (Model 2)
- Treatment With 3 Passes at 60 J/cm2: Single treatment with Liposonix System (Model 2) using grid repeat technique with 3 passes at 60 J/cm2 (180 J/cm2 total fluence)
  Liposonix System (Model 2)
Period: Overall Study
Arm/Group | Treatment at Level 1 | Treatment at Level 2 | Treatment at Level 3 | Treatment With 3 Passes at 60 J/cm2
Started | 18 | 20 | 17 | 17
Completed | 18 | 20 | 17 | 15
Not Completed | 0 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1
Not completed — Subject Noncompliance | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment at Level 1 | Treatment at Level 2 | Treatment at Level 3 | Treatment With 3 Passes at 60 J/cm2 | Total
Number analyzed (Participants) | 18 | 20 | 17 | 17 | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.4 (10.2) | 45.9 (12.3) | 42.4 (7.8) | 38.8 (10.9) | 43.0 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 15 | 16 | 16 | 64
  Male | 1 | 5 | 1 | 1 | 8
Region of Enrollment [Number; unit: participants]
  United States | 18 | 20 | 17 | 17 | 72
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 25.9 (2.4) | 25.2 (2.8) | 25.5 (2.8) | 25.4 (2.1) | 25.5 (2.5)

OUTCOME MEASURES:

1. Primary Outcome: Change in Waist Circumference 12 Weeks After Treatment as Compared to Baseline
Description: Change from baseline in waist circumference 12 weeks after treatment was assessed by blinded evaluators.
Time Frame: 12 weeks
Population: Intent-to-treat
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Treatment at Level 1 | Treatment at Level 2 | Treatment at Level 3 | Treatment With 3 Passes at 60 J/cm2
Number analyzed (Participants) | 18 | 20 | 17 | 17
cm | -1.6 (1.6) | -.96 (2.6) | -1.4 (2.4) | -1.2 (1.5)

2. Secondary Outcome: Change in Waist Circumference 4,8, and16 Weeks After Treatment as Compared to Baseline
Description: Change from baseline in waist circumference 4, 8, and 16 weeks after treatment was assessed by blinded evaluators.
Time Frame: 4 weeks, 8 weeks, 16 weeks
Population: Intent-to-treat
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Treatment at Level 1 | Treatment at Level 2 | Treatment at Level 3 | Treatment With 3 Passes at 60 J/cm2
Number analyzed (Participants) | 18 | 20 | 17 | 17
cm
  4 weeks | -0.66 (1.0) | -0.73 (1.6) | -0.86 (1.2) | -0.44 (0.9)
  8 weeks | -0.76 (1.3) | -1.3 (2.2) | -1.5 (1.7) | -0.92 (1.6)
  16 weeks | -1.8 (2.0) | -1.2 (3.0) | -1.4 (1.6) | -0.99 (2.0)

3. Secondary Outcome: Investigator Assessment of Improvement Using Global Aesthetic Improvement Scale (GAIS)
Description: GAIS evaluations were performed by Investigators at the 4, 8, 12, and 16 week visits. Investigators used direct visual assessment (live assessment) compared to photographs of subjects taken before treatment (baseline) to assess improvement in the treatment area.
  Scoring was based upon a five point grading System: 5 - Much Improved, 4 - Improved, 3 - No Change, 2 - Worse, or 1 - Much Worse. The definition of an improvement of the GAIS score included either a GAIS score of 'Improved' or 'Much Improved'.
Time Frame: 4, 8, 12, and 16 weeks
Population: Intent-to-treat
Measure: Number; unit: Percentage of subjects improved
Arm/Group | Treatment at Level 1 | Treatment at Level 2 | Treatment at Level 3 | Treatment With 3 Passes at 60 J/cm2
Number analyzed (Participants) | 18 | 20 | 17 | 17
Percentage of subjects improved
  4 weeks | 66.6 | 55.0 | 47.0 | 47.0
  8 weeks | 72.2 | 75.0 | 76.4 | 76.4
  12 weeks | 83.3 | 80.0 | 76.4 | 68.8
  16 weeks | 83.3 | 75.0 | 64.7 | 73.3

4. Secondary Outcome: Subject Assessment of Improvement Using Global Aesthetic Improvement Scale (GAIS)
Description: Subjects self-assessed improvement in the treatment area and assigned a GAIS score at each visit. Scoring was based upon a five point grading System: 5 - Much Improved, 4 - Improved, 3 - No Change, 2 - Worse, or 1 - Much Worse. The definition of an improvement of the GAIS score included either a GAIS score of 'Improved' or 'Much Improved'.
Time Frame: 4, 8, 12, and 16 weeks
Population: Intent-to-treat
Measure: Number; unit: percentage of subjects improved
Arm/Group | Treatment at Level 1 | Treatment at Level 2 | Treatment at Level 3 | Treatment With 3 Passes at 60 J/cm2
Number analyzed (Participants) | 18 | 20 | 17 | 17
percentage of subjects improved
  4 weeks | 77.7 | 55.0 | 52.9 | 52.9
  8 weeks | 61.1 | 84.2 | 70.5 | 76.4
  12 weeks | 72.2 | 100 | 68.8 | 75.0
  16 weeks | 77.7 | 75.0 | 64.7 | 73.3

5. Secondary Outcome: Subject Satisfaction With Treatment
Description: Subjects rated their satisfaction with treatment results using a 5-point Likert Satisfaction Scale (5: very satisfied; 4: satisfied; 3: neither satisfied nor dissatisfied; 2: dissatisfied; 1: very dissatisfied). The subject satisfaction score was analyzed as the proportion of subjects showing improvement as defined as a score of 4 or greater ('satisfied' or 'very satisfied').
Time Frame: 4, 8, 12, and 16 weeks
Population: Intent-to-treat
Measure: Number; unit: percentage of subjects satisfied
Arm/Group | Treatment at Level 1 | Treatment at Level 2 | Treatment at Level 3 | Treatment With 3 Passes at 60 J/cm2
Number analyzed (Participants) | 18 | 20 | 17 | 17
percentage of subjects satisfied
  4 weeks | 61.1 | 55.0 | 41.1 | 58.8
  8 weeks | 61.1 | 78.9 | 52.9 | 52.9
  12 weeks | 64.7 | 73.6 | 62.5 | 68.8
  16 weeks | 61.1 | 75.0 | 64.7 | 60.0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from day 0 through study exit
Arm/Group | Treatment at Level 1 | Treatment at Level 2 | Treatment at Level 3 | Treatment With 3 Passes at 60 J/cm2
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/20 | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 18/18 | 20/20 | 17/17 | 17/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment at Level 1 (N=18) | Treatment at Level 2 (N=20) | Treatment at Level 3 (N=17) | Treatment With 3 Passes at 60 J/cm2 (N=17)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea/vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (3)
Abdominal discomfort (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Burning sensation (General disorders) | 1 (1) | 2 (2) | 1 (1) | 2 (2)
Ecchymosis (General disorders) | 16 (16) | 20 (20) | 17 (18) | 16 (16)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain during treatment (General disorders) | 13 (13) | 13 (13) | 11 (11) | 10 (10)
Pain/tenderness (General disorders) | 17 (20) | 16 (19) | 16 (20) | 16 (20)
Paresthesia (General disorders) | 1 (1) | 1 (1) | 3 (3) | 2 (2)
Lumps/bumps (General disorders) | 3 (3) | 6 (6) | 1 (1) | 2 (2)
Soreness/discomfort (General disorders) | 0 (0) | 4 (4) | 1 (1) | 3 (3)
Swelling (General disorders) | 7 (7) | 8 (8) | 7 (7) | 7 (7)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Upper resp. tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infected arthropod bite (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bone fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Vasovagal episode (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chromaturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 5 (5) | 5 (5) | 5 (5) | 5 (5)
Erythema (Skin and subcutaneous tissue disorders) | 16 (16) | 14 (14) | 13 (13) | 12 (12)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Authorship and manuscript composition will reflect joint cooperation between the PI and Solta Medical personnel. Authorship will be established prior to the writing of the manuscript. No individual publications will be allowed prior to completion of the final report of the study except as agreed with Solta Medical. All publications must be reviewed and approved by Solta Medical prior to submission for publication.